CLINICAL TRIAL: NCT00793455
Title: Using Precision Performance Measurement To Conduct Focused Quality Improvement. Sub-Study 1.
Brief Title: Outreach for Patients With Uncompleted Colorectal Cancer Screening Orders
Acronym: UPQUAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kenzie Cameron, Research Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R18HS017163-01 (AHRQ)
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Results first posted 2011-12-01 (Estimated); Last update posted 2011-12-01 (Estimated); Status verified 2011-10

CONDITIONS: Colorectal Cancer Screening; Prevention & Control
Keywords: education; preventive service; screening

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Received Educational Outreach
  Interventions: Behavioral: Educational outreach
- Usual Care Control Group (No Intervention): Participants in this arm will receive normal care until outcome assessment is performed at 6 months following the placement of the order for the preventive service. They will be sent a letter reminding them to obtain the ordered preventive service test.

INTERVENTIONS:
Behavioral: Educational outreach — Participants will get a letter from their physician that explains that their records show the test has not been completed. The letter will be mailed along with an educational brochure and a DVD about colorectal cancer and colorectal cancer screening.
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to evaluate whether patient outreach is effective at increasing compliance with preventive screenings ordered by their physician. We hypothesize that educational outreach may increase completion rates.

DETAILED DESCRIPTION:
We designed an intervention to focus on patients who have received and accepted a referral for colonoscopy, yet have exhibited some barriers to screening as demonstrated by a lack of screening completion. We conducted a randomized controlled trial to assess the effects of a multicomponent intervention (patient reminder, print and multimedia materials) on colorectal screening completion among this target population.

ELIGIBILITY:
Inclusion Criteria:

* Patient's physician has ordered a preventive screening test
* Patient has not completed this test in 3 months
* Patient of Northwestern Medical Faculty Foundation General Internal Medicine Clinic.

Exclusion Criteria:

* Patient has been given a more recent order for the same screening test.
* Patient has significant life stress as noted in the Electronic Health Record (EHR)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 628 (Actual)
Dates: Start 2008-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenzie A Cameron, PhD, MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Medical Faculty Foundation General Internal Medicine Clinic, Chicago, Illinois, United States

REFERENCES:
- [Result] Cameron KA, Persell SD, Brown T, Thompson J, Baker DW. Patient outreach to promote colorectal cancer screening among patients with an expired order for colonoscopy: a randomized controlled trial. Arch Intern Med. 2011 Apr 11;171(7):642-6. doi: 10.1001/archinternmed.2010.468. Epub 2010 Dec 13. PMID 21149742

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial took place at a large urban academic primary care internal medicine practice in Chicago, IL. This trial was enrolling patients between October 2008 and May 2009.
Pre-assignment Details: We used data contained in the clinic's electronic health record to identify eligible patients. All eligible patients were randomly assigned in equal numbers to either the control or intervention arms. All eligible patients were randomized and assigned to groups until we reached target study size.
Groups:
- Intervention Group: Participants assigned to this group received a one-time educational intervention within one week of randomization. Educational intervention consisted of a letter from patient's physician, a brochure about colorectal cancer screening, and a DVD about colorectal cancer screening.
Period: Overall Study
Arm/Group | Intervention Group | Usual Care Control Group
Started | 314 | 314
Completed | 314 | 314
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Usual Care Control Group | Total
Number analyzed (Participants) | 314 | 314 | 628
Age Continuous [Mean (Standard Deviation); unit: years] | 57.90 (7.1) | 58.03 (6.6) | 58.0 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 197 | 192 | 389
  Male | 117 | 122 | 239
Race/Ethnicity, Customized [Number; unit: participants]
  White | 144 | 132 | 276
  Black | 79 | 77 | 156
  Hispanic | 9 | 14 | 23
  Other/unknown | 82 | 91 | 173
Region of Enrollment [Number; unit: participants]
  United States | 314 | 314 | 628
Number of visits in past 2 years [Number; unit: Participants]
  1-2 | 69 | 79 | 148
  3 | 80 | 79 | 159
  4 | 54 | 48 | 102
  >=5 | 111 | 108 | 219
Colorectal Cancer (CRC) screening history [Number; unit: Participants]
  Ever screened | 22 | 24 | 46
  Never screened | 292 | 290 | 582
Insurance Status [Number; unit: Participants]
  Private | 245 | 236 | 481
  Medicare | 56 | 63 | 119
  Medicaid | 10 | 10 | 20
  Uninsured | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Colorectal Cancer Screening Completion.
Description: We reviewed electronic health records of participants 3 months post randomization to ascertain outcome. We looked for one or both of the following (1) note in free text MD note documenting receipt of one form of colorectal cancer (CRC) screening during study period (2)lab results from fecal occult blood test, sigmoidoscopy, or colonoscopy.
  Participants were categorized as completing CRC screening if there was a lab result or physician note located in chart during study period. If no note or lab result was found in chart, then the participant was categorized as not completing CRC screening.
Time Frame: 3 months post randomization
Population: Analysis was based on intention to treat.
Measure: Number; unit: participants
Groups:
- Usual Care Control Group: Usual Care
Arm/Group | Usual Care Control Group | Intervention Group
Number analyzed (Participants) | 314 | 314
participants
  Did not Complete Screening | 304 | 283
  Completed Screening | 10 | 31
Statistical Analysis 1: Comparison: Usual Care Control Group vs Intervention Group; We compared the outcomes in the intervention and control groups using rate ratios and chi square test at 3 and 6 months, a 2 sided test with a p value < .05 was used to determine significance. The study was powered to detect a 10-percentage point difference in screening completion between intervention and control groups if the control rate of completion as 20% or less with 80% power; Test type: Superiority or Other; p < 0.05, Chi-squared; Rate Ratio = 3.1, 95% CI 2-sided [1.5 to 6.2]

2. Secondary Outcome: Colorectal Cancer Screening Completion
Description: We reviewed electronic health records of participants 6 months post randomization to ascertain outcome. We looked for one or both of the following (1) note in free text MD note documenting receipt of one form of colorectal cancer (CRC) screening during study period (2)lab results from fecal occult blood test, sigmoidoscopy, or colonoscopy.
  Participants were categorized as completing CRC screening if there was a lab result or physician note located in chart during study period. If no note or lab result was found in chart, then the participant was categorized as not completing CRC screening.
Time Frame: 6 months post randomization
Population: Analysis was based on intention to treat.
Measure: Number; unit: participants
Groups:
- Intervention Group: Received outreach intervention
Arm/Group | Usual Care Control Group | Intervention Group
Number analyzed (Participants) | 314 | 314
participants
  Completed Screening | 38 | 57
  Did not Complete Screening | 276 | 257
Statistical Analysis 1: Comparison: Usual Care Control Group vs Intervention Group; Same as primary outcome; Test type: Superiority or Other; p < 0.05, Chi-squared; Rate Ratio = 1.5, 95% CI 2-sided [1.03 to 2.2]

ADVERSE EVENTS:
Description: This was a minimal risk trial assessing an educational intervention which was approved by our Institutional Review Board with a waiver of consent. Serious and/or other adverse events were not collected or assessed.
Arm/Group | Intervention Group | Usual Care Control Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This study does not identify the timing of the intervention that would have the most impact. Mailings occurred 3 months or more after the order was placed, contacting patients sooner may have been more effective.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes